CLINICAL TRIAL: NCT04815486
Title: Clinical Effects of Immersive Multimodal BCI-VR Training After Bilateral Stimulation With rTMS on Upper Limb Motor Recovery After Stroke
Brief Title: Transcranial Magnetic Stimulation and Mental Representation Techniques for the Treatment of Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Collaborators: Hospital Beata María Ana (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Handboost
Record Dates: First submitted 2021-03-22; First posted 2021-03-25 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-03

CONDITIONS: Stroke
Keywords: Stroke; rTMS; Motor Imagery; BCI
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation; PUVA Therapy

STUDY DESIGN:
Intervention Model Description: The clinical trial will follow an AB/BA crossover design with a counterbalanced assignment, in which the first 50% of the sample will be assigned to order AB and the second 50% to order BA. The washout period between therapies A and B will be always a month.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilateral rTMS combined with MI through a BCI training platform in VR with NeuRow (Experimental): Sequential active rTMS at low frequency (healthy hemisphere) and high-frequency (injured hemisphere) application during 10 sessions in two weeks, and Motor Imagery (MI) treatment through the BCI training paradigm in VR (NeuRow) for 12 sessions in four weeks (3 sessions a week).The first 6 MI-neurofeedback sessions will carry out after bilateral stimulation with rTMS (i.e., rTMS as a priming method during the first two weeks), and the last 6 sessions, without rTMS as prior priming during the last two weeks
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Repetitive TMS in bilateral cortical primary motor area (Active Comparator): Sequential active rTMS at low frequency (healthy hemisphere) and high-frequency (injured hemisphere) application during 10 sessions in two weeks.
  Interventions: Device: Motor Imagery (MI) through a Brain-Computer Interface (BCI) training platform in Virtual Reality (VR) with NeuRow

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — Active rTMS in 10 daily sessions in two weeks of sequential application of: 90% RMT at 1Hz, 1000 pulses/day, 25s inter train on M1 of lesioned hemisphere and 90% RMT at 10Hz, 1000 pulses/day, 50s inter train on M1 of healthy hemisphere.
  Other Names: Therapy A
  Arms: Bilateral rTMS combined with MI through a BCI training platform in VR with NeuRow
Device: Motor Imagery (MI) through a Brain-Computer Interface (BCI) training platform in Virtual Reality (VR) with NeuRow — It will consist of a combination of the bilateral rTMS protocol and the MI-neurofeedback training. During this therapy, the patient received 10 consecutive daily sessions of bilateral rTMS (Monday to Friday, two weeks), with the same stimulation parameters as another therapy, and 12 non-consecutive sessions of MI-neurofeedback (three times a week for four weeks). The first 6 MI-neurofeedback sessions were carried out after bilateral stimulation with rTMS (i.e., rTMS as a priming method during the first two weeks), and the last 6 sessions, without rTMS as prior priming during the last two weeks.
  Other Names: Therapy B
  Arms: Repetitive TMS in bilateral cortical primary motor area

SUMMARY:
An immersive multimodal BCI-VR training and bilateral rTMS protocols are likely to complement their effects achieving a stronger neuroplasticity enhancement in stroke patients. Both have been used separately for the treatment of motor sequelae in the upper limbs after stroke. The main objective of this study is to carry out a double-blind, randomized, controlled trial aiming to study the clinical effect of Neurow system (NeuroRehabLab, Lisbon, Portugal) over bilateral rTMS plus conventional rehabilitation in upper limb motor sequelae after subacute stroke (3 to 12 months). We will look for changes in 1. Isometric strength in upper limb, 2. Functional motor scales of upper limb, 3. Hand dexterity 4. Cortical excitability changes. The investigators in the present project hypothesize that both neuromodulation techniques combined will be superior to the use of rTMS alone as adjuvant therapy to conventional rehabilitation.

DETAILED DESCRIPTION:
Stroke is a leading cause of long-term disability, it reduces mobility in more than half of stroke survivors age 65 and over.

Despite the lack of objective prognostic factors regarding the patient´s functionality after a stroke, we know that age, the level of initial disability, and the location and size of the lesion are elements that affect the evolution of post-stroke rehabilitation.

After stroke, the recovery of lost functions in the brain is achieved thanks to reorganizing networks in a process known as plasticity. Some damaged brain tissue may recover, or undamaged areas take over some functions.

One of the most relevant aspects of the rehabilitation prognosis is the time of evolution. After stroke, improvement is noticeably reduced over the second month, finding stabilization around the sixth month. One of the reasons for this is the reduction of neuroplasticity. There are indicative studies that reflect that, six months after a stroke, more than 60% of subjects will have a non-functional hand for Basic Activities of Daily Living (BADL), and 20-25% will not be able to walk without assistance. This determines the important global burden that stroke represents. It is relevant to emphasize the degree of disability after the rehabilitation process will be determined by the combination of existing motor, sensory and neuropsychological deficiencies.

In the last years, several non-invasive neuromodulation techniques have been shown efficient to enhance plasticity and stroke recovery. Among these interventions we can find exogenous neuromodulation, meaning that the neuromodulator stimulus comes from an external source, as is the case with rTMS (repetitive transcranial magnetic stimulation) which has the capacity to change the cortical excitability depending on the frequency of the magnetic pulses. Low frequencies (≤ 1 Hz) reduce local neural activity and high frequencies (≥ 5 Hz) increase cortical excitability. This technique has been successfully used bilaterally, stimulating the injured hemisphere and inhibiting the healthy one, to treat the interhemispheric inhibition phenomenon in stroke patients as it influences stroke recovery.

On the other hand, there are endogenous neuromodulation techniques that depend on the capacity of the subject to modulate its own brain activity. This can be achieved using neurofeedback (NFB), this consists of recording information of brain activity using electroencephalography (EEG) or functional magnetic resonance (fMRI) and displaying it to the subject in such way that he can receive a real time information of his own brain function. Virtual reality allows a new dimension on the neurofeedback immersion, and is likely to increase its efficacy. Stroke patients have been trained to reinforce certain EEG rhythms related with motor performance using NFB technique showing favourable effects on rehabilitation outcomes.

Some other techniques aiming to increase brain plasticity use the practice of imagination of movement of the affected hemibody. This is known as motor imagery and can be also enhanced through the use of brain computer interfaces. All the neuromodulation techniques are used to complement but not as a replacement of conventional rehabilitation.

On one hand exogenous neuromodulation effects are produced mainly by changes directly induced in cortical excitability and on the other hand endogenous neuromodulation is believed to have more widespread subcortical effects. One of the probable causes of the short-term effects of these techniques is the ceiling effect of changes in cortical excitability that can be achieved non-invasively, but despite of the good results achieved with the use of non-invasive neuromodulation techniques individually, there is a shortage of validated neurorehabilitation protocols that integrate different approaches that have been proven to be effective individually.

Neurow system (NeuroRehabLab, Lisbon, Portugal) is an immersive multimodal BCI-VR training system that combines motor imagery and neurofeedback through BCIs, using virtual reality has been designed to be used in chronic stroke patients, its efficacy has been shown in a pilot study.

Both approaches, the Neurow system (NeuroRehabLab, Lisbon, Portugal) and bilateral rTMS protocols are likely to complement their effects achieving a stronger neuroplasticity enhancement in stroke patients. Both have been used separately for the treatment of motor sequelae in the upper limbs after stroke. The effects of these combined techniques are not likely to be based only in the increase of cortical excitability but also on subcortical mechanisms.

The main objective of this study is to carry out a double-blind, randomized, controlled trial aiming to study the clinical effect of Neurow system (NeuroRehabLab, Lisbon, Portugal) over bilateral rTMS plus conventional rehabilitation in upper limb motor sequelae after subacute stroke (3 to 12 months). We will look for changes in 1. Isometric strength in upper limb, 2. Functional motor scales of upper limb, 3. Hand dexterity 4. Cortical excitability changes. Our main hypothesis is that both neuromodulation techniques combined will be superior to the use of rTMS alone as adjuvant therapy to conventional rehabilitation.

This protocol combines techniques that have proven to be cost-effective. If it is shown that the clinical improvement with this combination is significant, it will be open a new line of combined neuromodulation approaches to reach and effective method for the upper limb motor neurorehabilitation of after a stroke.

ELIGIBILITY:
Inclusion Criteria:

Older than 18 years old.

Ischemic or hemorrhagic cerebrovascular injury diagnosed by a neurologist and who have at least one brain-imaging test.

The onset of hemispheric ischemic or hemorrhagic stroke> 3 months.

Presence of upper limb motor sequelae due to stroke.

Sufficient cognitive ability to understand and perform tasks: Token Test> 11.

Stability in antispastic medication for more than 5 days.

Able to read and write.

Exclusion Criteria:

History of seizure or brain

Pacemakers, medication pumps, metal implants in the head (except dental implants)

Clinical unstability

Other pre-existing neurological diseases or previous cerebrovascular accidents with sequelae.

Sensory aphasia

Previous TMS after stroke

Hemispatial neglect,

Flaccid paralysis Brunnstrom's stage < 1

Visual problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Dynamometry | Baseline
  A handheld analogic dynamometer (Jamar® Plus+ Hand Dynamometer, 0-90 kg) will be used to assess isometric grip strength. Patients will be positioned in a straight back chair with both feet on the floor and the forearm resting on a stable surface. Each patient will be instructed to assume a position of adducted and neutrally rotated shoulder. For the arm to be tested, the elbow was flexed to 90º, the forearm and wrist will be in neutral positions, and the fingers will be flexed as needed for a maximal contraction. Patients will perform a maximal isometric grip contraction until they reach maximal force output. Three measures will be taken with 1-minute rest between test, and the mean value will be recorded
Change in Dynamometry | From Baseline at 2 weeks
  A handheld analogic dynamometer (Jamar® Plus+ Hand Dynamometer, 0-90 kg) will be used to assess isometric grip strength. Patients will be positioned in a straight back chair with both feet on the floor and the forearm resting on a stable surface. Each patient will be instructed to assume a position of adducted and neutrally rotated shoulder. For the arm to be tested, the elbow was flexed to 90º, the forearm and wrist will be in neutral positions, and the fingers will be flexed as needed for a maximal contraction. Patients will perform a maximal isometric grip contraction until they reach maximal force output. Three measures will be taken with 1-minute rest between test, and the mean value will be recorded
Change in Dynamometry | From Baseline at 4 weeks
  A handheld analogic dynamometer (Jamar® Plus+ Hand Dynamometer, 0-90 kg) will be used to assess isometric grip strength. Patients will be positioned in a straight back chair with both feet on the floor and the forearm resting on a stable surface. Each patient will be instructed to assume a position of adducted and neutrally rotated shoulder. For the arm to be tested, the elbow was flexed to 90º, the forearm and wrist will be in neutral positions, and the fingers will be flexed as needed for a maximal contraction. Patients will perform a maximal isometric grip contraction until they reach maximal force output. Three measures will be taken with 1-minute rest between test, and the mean value will be recorded
Change in Dynamometry | From Baseline at 6 weeks
  A handheld analogic dynamometer (Jamar® Plus+ Hand Dynamometer, 0-90 kg) will be used to assess isometric grip strength. Patients will be positioned in a straight back chair with both feet on the floor and the forearm resting on a stable surface. Each patient will be instructed to assume a position of adducted and neutrally rotated shoulder. For the arm to be tested, the elbow was flexed to 90º, the forearm and wrist will be in neutral positions, and the fingers will be flexed as needed for a maximal contraction. Patients will perform a maximal isometric grip contraction until they reach maximal force output. Three measures will be taken with 1-minute rest between test, and the mean value will be recorded
Change in Fugl-Meyer Assessment for upper extremity score | Baseline
  It is an observational rating scale that assesses sensorimotor impairments in post-stroke patients. It also includes four subscales: A. Upper Extremity (0-36), B. Wrist (0-10), C. Hand (0-14), D. Coordination/Speed (0-6) composing a total maximum score of 66 points. The therapist will rate each item according to direct observation of the motor performance, using a 3-point ordinal scale (0 = cannot perform, 1 = performs partially, and 2 = performs fully) with lower scores indicating more impairments. The FMA is easy to use and has excellent validity, reliability, and responsiveness.
Change in Fugl-Meyer Assessment for upper extremity score | From Baseline at 2 weeks
  It is an observational rating scale that assesses sensorimotor impairments in post-stroke patients. It also includes four subscales: A. Upper Extremity (0-36), B. Wrist (0-10), C. Hand (0-14), D. Coordination/Speed (0-6) composing a total maximum score of 66 points. The therapist will rate each item according to direct observation of the motor performance, using a 3-point ordinal scale (0 = cannot perform, 1 = performs partially, and 2 = performs fully) with lower scores indicating more impairments. The FMA is easy to use and has excellent validity, reliability, and responsiveness.
Change in Fugl-Meyer Assessment for upper extremity score | From Baseline at 4 weeks
  It is an observational rating scale that assesses sensorimotor impairments in post-stroke patients. It also includes four subscales: A. Upper Extremity (0-36), B. Wrist (0-10), C. Hand (0-14), D. Coordination/Speed (0-6) composing a total maximum score of 66 points. The therapist will rate each item according to direct observation of the motor performance, using a 3-point ordinal scale (0 = cannot perform, 1 = performs partially, and 2 = performs fully) with lower scores indicating more impairments. The FMA is easy to use and has excellent validity, reliability, and responsiveness.
Change in Fugl-Meyer Assessment for upper extremity score | From Baseline at 6 weeks
  It is an observational rating scale that assesses sensorimotor impairments in post-stroke patients. It also includes four subscales: A. Upper Extremity (0-36), B. Wrist (0-10), C. Hand (0-14), D. Coordination/Speed (0-6) composing a total maximum score of 66 points. The therapist will rate each item according to direct observation of the motor performance, using a 3-point ordinal scale (0 = cannot perform, 1 = performs partially, and 2 = performs fully) with lower scores indicating more impairments. The FMA is easy to use and has excellent validity, reliability, and responsiveness.
Change in Stroke Impact Scale score | Baseline
  It is a stroke-specific quality of life instrument to assess the consequences of stroke and to determine the quality of life improvement after stroke rehabilitation. It presents 4 subscales, but only hand function domain will be evaluated. Lower scores indicate more impairment in quality of life. The Minimal Detectable Change (MDC) and Clinically Important Difference (CID) of the hand function subscale are 25.9 and 17.8 points, respectively.
Change in Stroke Impact Scale score | From Baseline at 2 weeks
  It is a stroke-specific quality of life instrument to assess the consequences of stroke and to determine the quality of life improvement after stroke rehabilitation. It presents 4 subscales, but only hand function domain will be evaluated. Lower scores indicate more impairment in quality of life. The Minimal Detectable Change (MDC) and Clinically Important Difference (CID) of the hand function subscale are 25.9 and 17.8 points, respectively.
Change in Stroke Impact Scale score | From Baseline at 4 weeks
  It is a stroke-specific quality of life instrument to assess the consequences of stroke and to determine the quality of life improvement after stroke rehabilitation. It presents 4 subscales, but only hand function domain will be evaluated. Lower scores indicate more impairment in quality of life. The Minimal Detectable Change (MDC) and Clinically Important Difference (CID) of the hand function subscale are 25.9 and 17.8 points, respectively.
Change in Stroke Impact Scale score | From Baseline at 6 weeks
  It is a stroke-specific quality of life instrument to assess the consequences of stroke and to determine the quality of life improvement after stroke rehabilitation. It presents 4 subscales, but only hand function domain will be evaluated. Lower scores indicate more impairment in quality of life. The Minimal Detectable Change (MDC) and Clinically Important Difference (CID) of the hand function subscale are 25.9 and 17.8 points, respectively.
Change in Motricity Index of the Arm | Baseline
  The upper limb section of the MI assesses muscle strength in 3 muscle groups, including grip, elbow flexion, and shoulder separation. Each movement is scored discreetly (0 if there is no movement, 9 if the movement is palpable, 14 if the movement is visible, 19 if the movement is against gravity, 25 if the movement is against resistance and 33 if the movement is normal ), obtaining a total score for the upper limb that ranges from 0 (severely affected) to 100 (normal). This assessment methodology has been widely used in rehabilitation progress evaluation and counts with a normalized and weighted scoring system.
Change in Motricity Index of the Arm | From Baseline at 2 weeks
  The upper limb section of the MI assesses muscle strength in 3 muscle groups, including grip, elbow flexion, and shoulder separation. Each movement is scored discreetly (0 if there is no movement, 9 if the movement is palpable, 14 if the movement is visible, 19 if the movement is against gravity, 25 if the movement is against resistance and 33 if the movement is normal ), obtaining a total score for the upper limb that ranges from 0 (severely affected) to 100 (normal). This assessment methodology has been widely used in rehabilitation progress evaluation and counts with a normalized and weighted scoring system.
Change in Motricity Index of the Arm | From Baseline at 4 weeks
  The upper limb section of the MI assesses muscle strength in 3 muscle groups, including grip, elbow flexion, and shoulder separation. Each movement is scored discreetly (0 if there is no movement, 9 if the movement is palpable, 14 if the movement is visible, 19 if the movement is against gravity, 25 if the movement is against resistance and 33 if the movement is normal ), obtaining a total score for the upper limb that ranges from 0 (severely affected) to 100 (normal). This assessment methodology has been widely used in rehabilitation progress evaluation and counts with a normalized and weighted scoring system.
Change in Motricity Index of the Arm | From Baseline at 6 weeks
  The upper limb section of the MI assesses muscle strength in 3 muscle groups, including grip, elbow flexion, and shoulder separation. Each movement is scored discreetly (0 if there is no movement, 9 if the movement is palpable, 14 if the movement is visible, 19 if the movement is against gravity, 25 if the movement is against resistance and 33 if the movement is normal ), obtaining a total score for the upper limb that ranges from 0 (severely affected) to 100 (normal). This assessment methodology has been widely used in rehabilitation progress evaluation and counts with a normalized and weighted scoring system.

SECONDARY OUTCOMES:
Change in Electroencephalogram data | Baseline
  Mu (μ) is a type of rhythm in which α frequency can be found in sensorimotor cortex. Its changes are related with movement. M1 Mu (μ) rhythms will be assessed to evaluate changes in cortical function. They have been shown to be very useful in evaluating stroke patients recovery.
Change in Electroencephalogram data | At 2 weeks from Baseline
  Mu (μ) is a type of rhythm in which α frequency can be found in sensorimotor cortex. Its changes are related with movement. M1 Mu (μ) rhythms will be assessed to evaluate changes in cortical function. They have been shown to be very useful in evaluating stroke patients recovery.
Change in Electroencephalogram data | At 4 weeks from Baseline
  Mu (μ) is a type of rhythm in which α frequency can be found in sensorimotor cortex. Its changes are related with movement. M1 Mu (μ) rhythms will be assessed to evaluate changes in cortical function. They have been shown to be very useful in evaluating stroke patients recovery.
Change in Electroencephalogram data | At 6 weeks from Baseline
  Mu (μ) is a type of rhythm in which α frequency can be found in sensorimotor cortex. Its changes are related with movement. M1 Mu (μ) rhythms will be assessed to evaluate changes in cortical function. They have been shown to be very useful in evaluating stroke patients recovery.
Change in Nottingham Sensory Assessment (NSA) | Baseline
  Nottingham Sensory Assessment (NSA): Somatosensory impairment of the upper limb occurs in approximately 50% of adults after stroke, associated with loss of hand motor function, activity, and participation. The measurement of sensory impairment in the upper limb is a component of rehabilitation that contributes to the selection of sensorimotor techniques that optimize recovery and provide a prognostic estimate of the function of the affected upper limb.There are studies documenting changes produced in the sensation of the upper limb after the application of neurofeedback, and even after the intervention with motor imagery. Since the protocol presents an intervention with the application of these techniques, it is possible that there will be changes related to the sensitivity after the use of the platform, Neurow system (NeuroRehabLab, Lisbon, Portugal).
Change in Nottingham Sensory Assessment (NSA) | From Baseline at 4 weeks
  Nottingham Sensory Assessment (NSA): Somatosensory impairment of the upper limb occurs in approximately 50% of adults after stroke, associated with loss of hand motor function, activity, and participation. The measurement of sensory impairment in the upper limb is a component of rehabilitation that contributes to the selection of sensorimotor techniques that optimize recovery and provide a prognostic estimate of the function of the affected upper limb.There are studies documenting changes produced in the sensation of the upper limb after the application of neurofeedback, and even after the intervention with motor imagery. Since the protocol presents an intervention with the application of these techniques, it is possible that there will be changes related to the sensitivity after the use of the platform, Neurow system (NeuroRehabLab, Lisbon, Portugal).
Change in Nottingham Sensory Assessment (NSA) | From Baseline at 6 weeks
  Nottingham Sensory Assessment (NSA): Somatosensory impairment of the upper limb occurs in approximately 50% of adults after stroke, associated with loss of hand motor function, activity, and participation. The measurement of sensory impairment in the upper limb is a component of rehabilitation that contributes to the selection of sensorimotor techniques that optimize recovery and provide a prognostic estimate of the function of the affected upper limb.There are studies documenting changes produced in the sensation of the upper limb after the application of neurofeedback, and even after the intervention with motor imagery. Since the protocol presents an intervention with the application of these techniques, it is possible that there will be changes related to the sensitivity after the use of the platform, Neurow system (NeuroRehabLab, Lisbon, Portugal).
Change in Finger Tapping Task | Baseline
  It measures motor function and is very sensitive to the slowing down of responses. In this task, following the Strauss application norms, the participants will be instructed to press the space-bar on the keyboard as fast as possible and repeatedly with the index finger. Five 10-second attempts will be performed with the dominant hand. The average time between two consecutive taps in the five trials will be the dependent variable.
Change in Finger Tapping Task | From Baseline at 4 weeks
  It measures motor function and is very sensitive to the slowing down of responses. In this task, following the Strauss application norms, the participants will be instructed to press the space-bar on the keyboard as fast as possible and repeatedly with the index finger. Five 10-second attempts will be performed with the dominant hand. The average time between two consecutive taps in the five trials will be the dependent variable.
Change in Finger Tapping Task | From Baseline at 6 weeks
  It measures motor function and is very sensitive to the slowing down of responses. In this task, following the Strauss application norms, the participants will be instructed to press the space-bar on the keyboard as fast as possible and repeatedly with the index finger. Five 10-second attempts will be performed with the dominant hand. The average time between two consecutive taps in the five trials will be the dependent variable.
Change in Nine Hole Peg Test | Baseline
  It evaluates the impairment in upper limb dexterity. Patients must pick up as quick as possible, nine pegs from a container one-by-one unimanually and transfer them into a target pegboard with nine holes until filled. Then, they must return them unimanually to the container. The outcome variable will be the time spent to complete the whole task. This test is considered reliable, valid, and sensitive to change, among stroke patients.
Change in Nine Hole Peg Test | From Baseline at 4 weeks
  It evaluates the impairment in upper limb dexterity. Patients must pick up as quick as possible, nine pegs from a container one-by-one unimanually and transfer them into a target pegboard with nine holes until filled. Then, they must return them unimanually to the container. The outcome variable will be the time spent to complete the whole task. This test is considered reliable, valid, and sensitive to change, among stroke patients.
Change in Nine Hole Peg Test | From Baseline at 6 weeks
  It evaluates the impairment in upper limb dexterity. Patients must pick up as quick as possible, nine pegs from a container one-by-one unimanually and transfer them into a target pegboard with nine holes until filled. Then, they must return them unimanually to the container. The outcome variable will be the time spent to complete the whole task. This test is considered reliable, valid, and sensitive to change, among stroke patients.
Change in Modified Ashworth Scale score | Baseline
  Patients will be in the supine position with their arms by their side and with their head in neutral position. Wrist and elbow muscles resistance will be assessed during two repetitions of a passive motion within one second and measured on the following scale: 0 = no increased resistance; 1 = slightly increase resistance (at the end of the range of motion); 1+ = slightly increase resistance (less than half of the range of motion); 2 = clear resistance (most of the range of motion); 3 = strong resistance; 4 = rigid flexion or extension. It is markedly responsive in detecting the changes in muscle tone in patients with stroke and its minimal clinically important difference of effect sizes 0.5 and 0.8 standard deviations for the upper extremity muscles are 0.48 and 0.76, respectively.
Change in Modified Ashworth Scale score | Baseline at 4 weeks
  Patients will be in the supine position with their arms by their side and with their head in neutral position. Wrist and elbow muscles resistance will be assessed during two repetitions of a passive motion within one second and measured on the following scale: 0 = no increased resistance; 1 = slightly increase resistance (at the end of the range of motion); 1+ = slightly increase resistance (less than half of the range of motion); 2 = clear resistance (most of the range of motion); 3 = strong resistance; 4 = rigid flexion or extension. It is markedly responsive in detecting the changes in muscle tone in patients with stroke and its minimal clinically important difference of effect sizes 0.5 and 0.8 standard deviations for the upper extremity muscles are 0.48 and 0.76, respectively.
Change in Modified Ashworth Scale score | Baseline at 6 weeks
  Patients will be in the supine position with their arms by their side and with their head in neutral position. Wrist and elbow muscles resistance will be assessed during two repetitions of a passive motion within one second and measured on the following scale: 0 = no increased resistance; 1 = slightly increase resistance (at the end of the range of motion); 1+ = slightly increase resistance (less than half of the range of motion); 2 = clear resistance (most of the range of motion); 3 = strong resistance; 4 = rigid flexion or extension. It is markedly responsive in detecting the changes in muscle tone in patients with stroke and its minimal clinically important difference of effect sizes 0.5 and 0.8 standard deviations for the upper extremity muscles are 0.48 and 0.76, respectively.
Change in TMS Resting Motor Threshold (RMT) and cortical silent period (CSP) | Baseline
  In the first dorsal interosseous muscle or the abductor pollicis brevis muscle will be recorded to determine the cortical excitability changes and correlate them with the clinical outcomes.
Change in TMS Resting Motor Threshold (RMT)and cortical silent period (CSP) | From Baseline at 2 weeks
  In the first dorsal interosseous muscle or the abductor pollicis brevis muscle will be recorded to determine the cortical excitability changes and correlate them with the clinical outcomes.
Change in TMS Resting Motor Threshold (RMT)and cortical silent period (CSP) | From Baseline at 4 weeks
  In the first dorsal interosseous muscle or the abductor pollicis brevis muscle will be recorded to determine the cortical excitability changes and correlate them with the clinical outcomes.
Change in TMS Resting Motor Threshold (RMT) and cortical silent period (CSP) | From Baseline at 6 weeks
  In the first dorsal interosseous muscle or the abductor pollicis brevis muscle will be recorded to determine the cortical excitability changes and correlate them with the clinical outcomes.
Change in Barthel Index(BI) | Baseline
  Accurately assessing the ADLs of stroke patients greatly helps in evaluating the efficacy of stroke treatments. The Barthel Index was originally established to assess ADL in stroke patients and has been used extensively for this purpose.
Change in Barthel Index(BI) | From Baseline at 4 weeks
  Accurately assessing the ADLs of stroke patients greatly helps in evaluating the efficacy of stroke treatments. The Barthel Index was originally established to assess ADL in stroke patients and has been used extensively for this purpose.
Change in Barthel Index(BI) | From Baseline at 6 weeks
  Accurately assessing the ADLs of stroke patients greatly helps in evaluating the efficacy of stroke treatments. The Barthel Index was originally established to assess ADL in stroke patients and has been used extensively for this purpose.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Pablo Romero Muñoz, MD PhD, Principal Investigator — Universidad Francisco de Vitoria, Facultad de Ciencias Experimentales
Locations (1):
- Hospital Beata Maria Ana, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual anonymized participant data will be available to other researchers under request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Six months at the end of the study.
Access Criteria: Individual anonymized participant data will be available to other researchers under request.

REFERENCES:
- [Background] Vourvopoulos A, Bermudez I Badia S. Motor priming in virtual reality can augment motor-imagery training efficacy in restorative brain-computer interaction: a within-subject analysis. J Neuroeng Rehabil. 2016 Aug 9;13(1):69. doi: 10.1186/s12984-016-0173-2. PMID 27503007
- [Background] Vourvopoulos A, Jorge C, Abreu R, Figueiredo P, Fernandes JC, Bermudez I Badia S. Efficacy and Brain Imaging Correlates of an Immersive Motor Imagery BCI-Driven VR System for Upper Limb Motor Rehabilitation: A Clinical Case Report. Front Hum Neurosci. 2019 Jul 11;13:244. doi: 10.3389/fnhum.2019.00244. eCollection 2019. PMID 31354460
- [Background] Takeuchi N, Izumi S. Maladaptive plasticity for motor recovery after stroke: mechanisms and approaches. Neural Plast. 2012;2012:359728. doi: 10.1155/2012/359728. Epub 2012 Jun 26. PMID 22792492
- [Background] Takeuchi N, Tada T, Toshima M, Matsuo Y, Ikoma K. Repetitive transcranial magnetic stimulation over bilateral hemispheres enhances motor function and training effect of paretic hand in patients after stroke. J Rehabil Med. 2009 Nov;41(13):1049-54. doi: 10.2340/16501977-0454. PMID 19894000
- [Background] Zhang L, Xing G, Shuai S, Guo Z, Chen H, McClure MA, Chen X, Mu Q. Low-Frequency Repetitive Transcranial Magnetic Stimulation for Stroke-Induced Upper Limb Motor Deficit: A Meta-Analysis. Neural Plast. 2017;2017:2758097. doi: 10.1155/2017/2758097. Epub 2017 Dec 21. PMID 29435371
- [Background] Pichiorri F, Morone G, Petti M, Toppi J, Pisotta I, Molinari M, Paolucci S, Inghilleri M, Astolfi L, Cincotti F, Mattia D. Brain-computer interface boosts motor imagery practice during stroke recovery. Ann Neurol. 2015 May;77(5):851-65. doi: 10.1002/ana.24390. Epub 2015 Mar 27. PMID 25712802
- [Background] Dionisio A, Duarte IC, Patricio M, Castelo-Branco M. The Use of Repetitive Transcranial Magnetic Stimulation for Stroke Rehabilitation: A Systematic Review. J Stroke Cerebrovasc Dis. 2018 Jan;27(1):1-31. doi: 10.1016/j.jstrokecerebrovasdis.2017.09.008. Epub 2017 Oct 27. PMID 29111342
- [Background] Sasaki N, Mizutani S, Kakuda W, Abo M. Comparison of the effects of high- and low-frequency repetitive transcranial magnetic stimulation on upper limb hemiparesis in the early phase of stroke. J Stroke Cerebrovasc Dis. 2013 May;22(4):413-8. doi: 10.1016/j.jstrokecerebrovasdis.2011.10.004. Epub 2011 Dec 15. PMID 22177936
- [Background] Pfurtscheller G, Neuper C, Muller GR, Obermaier B, Krausz G, Schlogl A, Scherer R, Graimann B, Keinrath C, Skliris D, Wortz M, Supp G, Schrank C. Graz-BCI: state of the art and clinical applications. IEEE Trans Neural Syst Rehabil Eng. 2003 Jun;11(2):177-80. doi: 10.1109/TNSRE.2003.814454. PMID 12899267
- [Background] Cogne M, Gil-Jardine C, Joseph PA, Guehl D, Glize B. Seizure induced by repetitive transcranial magnetic stimulation for central pain: Adapted guidelines for post-stroke patients. Brain Stimul. 2017 Jul-Aug;10(4):862-864. doi: 10.1016/j.brs.2017.03.010. Epub 2017 Mar 23. No abstract available. PMID 28359831
- [Background] Duncan PW, Wallace D, Lai SM, Johnson D, Embretson S, Laster LJ. The stroke impact scale version 2.0. Evaluation of reliability, validity, and sensitivity to change. Stroke. 1999 Oct;30(10):2131-40. doi: 10.1161/01.str.30.10.2131. PMID 10512918